CLINICAL TRIAL: NCT03843307
Title: Study to Evaluate the Tennant Biomodulator® PRO Device Designed by AVAZZIA Effects on Perfusion
Brief Title: Avazzia-University of Texas Southwestern Medical Center-Tennant Biomodulator® PRO Perfusion Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties with enrollment which were complicated by pauses to clinical research from COVID, The University of Texas Southwestern has decided not to pursue the continuation of this study.
Sponsor: Avazzia, Inc (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other); Lawrence A. Lavery, DPM, MPH (Unknown); Kathryn Davis, Ph.D. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 042018-005
Record Dates: First submitted 2019-02-07; First posted 2019-02-18 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Perfusion; Complications; Wound; Foot
Keywords: Electrical stimulation; Perfusion; Foot wound; Foot pain
MeSH Terms: conditions — Foot Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Electrical stimulation (Experimental)
  Interventions: Device: Avazzia Tennant Biomodulator® PRO

INTERVENTIONS:
Device: Avazzia Tennant Biomodulator® PRO — High-voltage pulsed current (HVPC) electrical stimulation with Reactions and BEST™ (Bio-Electric Stimulation Technology) microcurrent that measure and change with tissue electrical characteristics.

SUMMARY:
This study is an open label trial designed to test the effectiveness of the Tennant Biomodulator® PRO electrical stimulation device (Avazzia), which uses BEST™ (Bio-Electric Stimulation Technology), on hospital in-patients to improve perfusion in the treated and contralateral limb.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide Informed Consent
* Ankle Brachial Index (ABI) ≥ 0.5 (bedside ABI is acceptable for screening purposes as the formal imaging ABI may not be resulted prior to therapy)
* Participant is a hospital in-patient for the duration of study procedures
* One or more chronic lower extremity wounds that are located in the ankle area or below that has persisted a minimum of 30 days prior to the Screening visit
* 18 years of age or older

Exclusion Criteria:

* Unable to provide informed consent
* <18 years of age
* Participant has a demand-type cardiac pacemaker, implanted defibrillator or other implanted metallic or electronic device.
* Participant has untreated osteomyelitis
* Participant has active cellulitis
* Participant has active charcot
* Is pregnant or plans to become pregnant
* Is nursing or actively lactating
* Developmental disability/significant psychological disorder that in the opinion of the investigator could impair the participant's ability to provide informed consent, participate in the study protocol including untreated schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Improvement in perfusion up to 3 hours | 3 hours
  Change in skin perfusion will be assessed by Skin Perfusion Pressure Test (SPP)
Improvement in perfusion up to 3 hours | 3 hours
  Change in skin perfusion will be assessed by Hyperspectral Imaging (HSI)

SECONDARY OUTCOMES:
Duration of BEST-induced perfusion effects | 3 hours
  To compare the duration of BEST™ (Bio-Electric Stimulation Technology) induced perfusion effects
Changes in reported pain after BEST™ (Bio-Electric Stimulation Technology) administration, at the point perfusion returns to baseline, and at 24 hours after treatment | 24 hours
  Pain will be assessed with the Visual Analog Scale (VAS) labeled from '0': no pain to '10': worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM, MPH, Principal Investigator — University of Texas Southwestern Medical Center, Department of Plastic Surgery
Locations (1):
- University of Texas Southwestern Medical Center, Department of Plastic Surgery, Dallas, Texas, United States

REFERENCES:
- [Background] Thakral G, Lafontaine J, Najafi B, Talal TK, Kim P, Lavery LA. Electrical stimulation to accelerate wound healing. Diabet Foot Ankle. 2013 Sep 16;4. doi: 10.3402/dfa.v4i0.22081. PMID 24049559
- [Background] Peters EJ, Armstrong DG, Wunderlich RP, Bosma J, Stacpoole-Shea S, Lavery LA. The benefit of electrical stimulation to enhance perfusion in persons with diabetes mellitus. J Foot Ankle Surg. 1998 Sep-Oct;37(5):396-400; discussion 447-8. doi: 10.1016/s1067-2516(98)80048-3. PMID 9798171
- [Background] Nair HKR. Microcurrent as an adjunct therapy to accelerate chronic wound healing and reduce patient pain. J Wound Care. 2018 May 2;27(5):296-306. doi: 10.12968/jowc.2018.27.5.296. PMID 29738296
- [Background] Andrushko JW, Lanovaz JL, Bjorkman KM, Kontulainen SA, Farthing JP. Unilateral strength training leads to muscle-specific sparing effects during opposite homologous limb immobilization. J Appl Physiol (1985). 2018 Apr 1;124(4):866-876. doi: 10.1152/japplphysiol.00971.2017. Epub 2017 Dec 14. PMID 29357520